CLINICAL TRIAL: NCT00823264
Title: Prospective Randomized Study of Multidose Activated Charcoal in Supratherapeutic Phenytoin Serum Levels
Brief Title: Phenytoin and Multidose Activated Charcoal
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Emory University (Other)
Responsible Party: Principal Investigator, Brent W Morgan, MD, Associate Professor, Emory University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB00008017
Record Dates: First submitted 2009-01-14; First posted 2009-01-15 (Estimated); Results first posted 2014-09-11 (Estimated); Last update posted 2014-09-11 (Estimated); Status verified 2014-09

CONDITIONS: Phenytoin Toxicity
Keywords: Anticonvulsants; Toxicology; multidose charcoal; phenytoin
MeSH Terms: interventions — Charcoal

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Multiple Doses of Activated Charcoal (Experimental): Patients will receive 50 grams of activated charcoal by mouth every 4 hours until phenytoin levels drop below 25 ug/cc
  Interventions: Drug: Activated Charcoal
- Control (No Intervention): Will not receive activated charcoal. Serum levels will be followed.

INTERVENTIONS:
Drug: Activated Charcoal — 50 grams by mouth every 4 hours until serum phenytoin level is less than 25.
  Other Names: Charcoal
  Arms: Multiple Doses of Activated Charcoal

SUMMARY:
Phenytoin is a medicine used to treat seizures. If too much is taken, patients have ill effects including sleepiness, unsteady gait, and eye problems. The amount of drug in their system can be measured in their blood. Charcoal is a medicine that can absorb phenytoin. We want to see if giving multiple doses of charcoal will quicken the removal of phenytoin from the blood. This is theorized to occur as charcoal absorbs phenytoin from across the intestines and then is secreted in the stool. Patients will be selected to receive either charcoal in multiple doses or no charcoal and their serum levels will be drawn repeatedly to follow their level. The different groups will then be compared to see if multidose charcoal does indeed increase the elimination of phenytoin from the body.

DETAILED DESCRIPTION:
See above

ELIGIBILITY:
Inclusion Criteria:

* Phenytoin level > 30 mg/L

Exclusion Criteria:

* Age < 18
* Known allergy to Activated Charcoal
* Pregnant
* Inability to take PO drugs
* Non English speaking
* Inability to give consent
* Any prisoners

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2008-08; Primary Completion 2010-07 (Actual); Study Completion 2012-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Carl Skinner, MD, Principal Investigator — Emory University
Locations (1):
- Grady Memorial Hospital, Atlanta, Georgia, United States

REFERENCES:
- [Result] Skinner CG, Chang AS, Matthews AS, Reedy SJ, Morgan BW. Randomized controlled study on the use of multiple-dose activated charcoal in patients with supratherapeutic phenytoin levels. Clin Toxicol (Phila). 2012 Sep;50(8):764-9. doi: 10.3109/15563650.2012.716159. Epub 2012 Aug 17. PMID 22897408

RESULTS

PARTICIPANT FLOW:
Groups:
- Multiple Doses of Activated Charcoal: Will receive 50 grams of activated charcoal every 4 hours by mouth until phenytoin level is < 25 ug/cc.
Period: Overall Study
Arm/Group | Control | Multiple Doses of Activated Charcoal
Started | 10 | 7
Completed | 8 | 7
Not Completed | 2 | 0
Not completed — Protocol Violation | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- Multiple Doses of Activated Charcoal: Will receive 50 grams of activated charcoal by mouth every 4 hours until phenytoin levels are < 25 ug/cc.
- Total: Total of all reporting groups
Arm/Group | Control | Multiple Doses of Activated Charcoal | Total
Number analyzed (Participants) | 8 | 7 | 15
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 7 | 7 | 14
  >=65 years | 1 | 0 | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 8 | 7 | 15
Region of Enrollment [Number; unit: participants]
  United States | 8 | 7 | 15

OUTCOME MEASURES:

1. Primary Outcome: Time of Elimination of Phenytoin in Patients With Elevated Phenytoin Levels
Description: We enrolled patients with elevated phenytoin levels into the study with greater than 30 ug/cc. The treatment arm received multiple doses of activated charcoal and the control arm received no activated charcoal. We obtained serum phenytoin levels every 6 hours for 24 hours then once every 24 hours. The time to reach a subtoxic level was determined in each arm by looking at serum phenytoin levels and documenting when it was below 25 ug/cc.
Time Frame: Serum phenytoin levels were obtained every 6 hours for 24 hours then once every 24 hours
Measure: Median (Inter-Quartile Range); unit: hours
Groups:
- Multiple Doses of Activated Charcoal: Patients received 50 grams of activated charcoal by mouth every 6 hours until the phenytoin levels was below 25 ug/cc.
Arm/Group | Control | Multiple Doses of Activated Charcoal
Number analyzed (Participants) | 8 | 7
hours | 41.1 [11.6 to 196] | 19.3 [13 to 33]
Statistical Analysis 1: Comparison: Control vs Multiple Doses of Activated Charcoal; Test type: Superiority or Other; p = 0.049, Wilcoxon (Mann-Whitney)

ADVERSE EVENTS:
Time Frame: Participants were followed for the duration of hospital stay, an average of 24 hours
Groups:
- Multiple Doses of Charcoal: Patients received 50 grams of activated charcoal by mouth every 6 hours until the phenytoin levels was below 25 ug/cc.
Arm/Group | Multiple Doses of Charcoal | Control
Serious Adverse Events (participants affected / at risk) | 0/7 | 0/8
Other Adverse Events (participants affected / at risk) | 0/7 | 0/8

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes